CLINICAL TRIAL: NCT04419688
Title: A Double-blind, Randomised, Placebo-controlled, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple-ascending Doses of Intravenously Administered STT-5058 in Otherwise Healthy Subjects With Elevated Triglyceride Levels and Single-ascending and Multiple Doses of Subcutaneously Administered STT-5058 in Otherwise Healthy Subjects With Elevated Triglyceride Levels and Patient Volunteers With Hypertriglyceridemia.
Brief Title: A First in Human Study of STT-5058, an Antibody That Binds ApoC3
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: recruitment failure
Sponsor: Staten Biotechnology BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STT-01
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STT-5058 (Experimental)
  Interventions: Drug: STT-5058
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STT-5058 — Monoclonal Antibody STT-5058
  Arms: STT-5058
Drug: Placebo — Matching placebo to STT-5058
  Arms: Placebo

SUMMARY:
A First in Human Study of STT-5058, an Antibody That Binds ApoC3, investigating single and multiple ascending intravenous doses and ascending subcutaneous doses of STT-5058 in otherwise healthy volunteers with elevated triglyceride levels

DETAILED DESCRIPTION:
The study is in five parts. Part A is up to 6 single ascending intravenous dose cohorts of STT-5058 in otherwise healthy volunteers with TRGs >150mg/dL. Part B is up to 4 multiple ascending intravenous dose cohorts of STT-5058 in otherwise healthy volunteers with TRGs >150mg/dL who will receive 3 doses at 2 week intervals. Part C will recruit a single cohort of patient volunteers with TRG >200mg/dL who will receive 3 doses at 2 week intervals of STT-5058. Part D will investigate up to 2 single ascending doses of subcutaneous STT-5058. Part E will recruit a single cohort of otherwise healthy volunteers with TRG > 150mg/dL to receive 4 doses subcutaneously of STT-5058 over 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* in good health
* Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception Parts A, B and D
* BMI between 18 and 35 kg/m2 inclusive
* Fasting Triglycerides between 150 and 400mg/dL inclusive Part C
* Fasting Triglycerides between 200 and 400 mg/dL inclusive
* Fasting LDL-C between 70 and 160 mg/dL inclusive
* BMI between 18 and 40 kg/m2

Exclusion Criteria:

* significant history or clinical manifestation of metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator
* Confirmed (eg, 2 consecutive measurements) systolic blood pressure >150 or <90 mmHg, diastolic blood pressure >90 or <50 mmHg, and heart rate >90 or <40 beats per minute at Screening, Check-in, or prior to dosing on Day 1.
* History of alcoholism or drug/chemical abuse within 2 years prior to Check-in.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days or 5 half-lives (if known), whichever is longer, prior to dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 10 weeks
  incidence and severity of adverse events

SECONDARY OUTCOMES:
AUC | 10-14 weeks
  Area under the PK curve
Cmax | 24 hours
  Maximum concentration
Half life | 10-14 weeks
  time to reduction in plasma levels by 50%

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Leeds Clinical Research Unit, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No